CLINICAL TRIAL: NCT02611596
Title: Does Ranolazine Decrease Biomarkers That Indicate Evidence of Myocardial Damage in Diabetics With Stable Ischemic Heart Disease? A Double-blinded, Randomized, Placebo Controlled Trial
Brief Title: Does Ranolazine Decrease Biomarkers of Myocardial Damage in Diabetics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Todd C. Villines, MD, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 409189
Record Dates: First submitted 2015-11-18; First posted 2015-11-23 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Silent Myocardial Ischemia; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine (Experimental): Subjects will take one 500mg tablet twice daily (500mg BID) for seven days and then increase to two 500mg tablets twice daily (1000mg BID) for the remainder of the study, for a total of 24 weeks. Subjects taking moderate CYP3A4 inhibitors will not participate in upward titration and will remain on 500mg tablet twice daily (500mg BID) for the duration of the trial.
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Subjects will take one placebo tablet (identical to the 500mg Ranolazine tablet) twice daily (500mg BID) for seven days and then increase to two 500mg tablets twice daily (1000mg BID) for the remainder of the study, for a total of 24 weeks. Subjects taking moderate CYP3A4 inhibitors will not participate in upward titration and will remain on 500mg tablet twice daily (500mg BID) for the duration of the trial.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — 24 weeks of the assigned medication
  Arms: Ranolazine
Drug: Placebo — Placebo for 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this investigation is to compare subjects at high risk for silent myocardial ischemia in the placebo group to subjects at high risk for silent myocardial ischemia in the ranolazine group to determine if ranolazine can be used as a treatment to decrease silent myocardial ischemia (SMI). Subjects at high risk for silent myocardial ischemia are defined in this protocol as diabetics with stable ischemic heart disease. This study will look at the impact ranolazine treatment has on biomarkers that have been shown to be highly associated with increased risk of morbidity and mortality in relation to SMI. If the hypothesis is correct, further studies can be conducted to determine if treatment with ranolazine has impact on long-term outcomes such as hospitalizations, myocardial infarction, congestive heart failure or sudden cardiac death.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at risk for silent myocardial ischemia as defined by:
* Stable ischemic heart disease as defined by:

  * Obstruction of at least one epicardial vessel of > 50 percent by invasive or non-invasive coronary angiography, or
  * Evidence of ischemia or infarct on SPECT imaging, or
  * History of myocardial infarction > 3 months ago, or
  * Stent placement (PCI) > 3 months ago, or
  * Coronary artery bypass grafting (CABG) > 3 months ago AND
* Type 2 diabetics as defined by:

  * HgbA1C ≥ 6.5 percent, or
  * Fasting Blood Glucose > 125 mg/dL on two or more blood draws, or
  * Random Blood Glucose of ≥ 200 mg/dL on a single blood draw, or
  * Previous diagnosis of type 2 diabetes listed in the subject's medical record AND

    - On Optimal Medical Therapy as defined as being on ALL of the following at time of enrollment:
  * Beta Blocker
  * Aspirin
  * Statin AND
* Females < 60 who have not been free of menstruation for 2 years (menopause diagnosed) or who do not have documented history of hysterectomy must be willing to use at least one form of birth control (including abstinence as an option) for the duration of the study. If condoms are the method chosen, they are strongly urged to use a second form of birth control in addition to condoms.

AND

Screening Criteria met:

• hs cTnT > 0.014 ng/mL

Exclusion Criteria:

* Percutaneous intervention/stent placement in the past 3 months
* Coronary artery bypass grafting in the past 3 months
* Treatment with ranolazine in the past 12 months
* Significant lung disease, COPD or use of supplemental oxygen
* Cirrhosis
* Estimated Glomerular Filtration Rate (GFR) < 30
* Subject taking strong CYP3A inhibitors (ketoconazole, itraconazole, clarithryomycin, nefazodone, nelfinavir, ritonavir, indinavir and saquinavir)
* Subject taking strong CYP3A inducers (rifampin, rifabutin, rifapentin, phenobarbital, phenytoin, carbamazepine, St. John's wort)
* Subjects taking P-gp Inhibitors (cyclosporine)
* Subject is taking concurrent simvastatin in > 20 mg/day
* Subject is taking metformin > 1700 mg/day
* NYHA Class 3 or 4 Heart Failure (severe)
* Canadian Cardiovascular Society Grade 4 Angina
* Unstable angina defined as a new angina occurring after minimal exercise or at rest OR a significant increase in angina severity (≥ 2 CCS grades) occurring with minimal exertion, with high clinical suspicion of acute coronary syndrome.
* Planned PCI or Cardiac Surgery
* Pregnant females or females trying to become pregnant
* Breast-feeding females
* Subjects younger than age 30 or older than age 85
* Lactose Intolerance (placebo has lactose monohydrate)
* Lactose/Milk allergy (placebo has lactose monohydrate)
* QTc > 500 msec

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
hs cTnT | 24 weeks
  Does ranolazine decrease hs cTnT in subjects at high risk for silent myocardial ischemia?
NT-pro-BNP | 24 weeks
  Does ranolazine decrease NT-pro-BNP in subjects at high risk for silent myocardial ischemia?
hsCRP | 24 weeks
  Determine the degree of decrease of hs CRP in subjects in the ranolazine group.

SECONDARY OUTCOMES:
prevalence of hs cTnT > 99th percentile | 24 weeks
  Determine the prevalence of hs cTnT greater than the 99th percentile (0.014 ng/mL) in asymptomatic diabetic subjects with stable ischemic heart disease.

CONTACTS AND LOCATIONS:
Overall Officials: Todd C Villines, MD, Principal Investigator — WRNMMC

REFERENCES:
- [Background] Marzilli M, Merz CN, Boden WE, Bonow RO, Capozza PG, Chilian WM, DeMaria AN, Guarini G, Huqi A, Morrone D, Patel MR, Weintraub WS. Obstructive coronary atherosclerosis and ischemic heart disease: an elusive link! J Am Coll Cardiol. 2012 Sep 11;60(11):951-6. doi: 10.1016/j.jacc.2012.02.082. PMID 22954239
- [Background] Cannon RO 3rd. Microvascular angina and the continuing dilemma of chest pain with normal coronary angiograms. J Am Coll Cardiol. 2009 Sep 1;54(10):877-85. doi: 10.1016/j.jacc.2009.03.080. PMID 19712795
- [Background] Deedwania PC, Carbajal EV. Silent ischemia during daily life is an independent predictor of mortality in stable angina. Circulation. 1990 Mar;81(3):748-56. doi: 10.1161/01.cir.81.3.748. PMID 2306826
- [Background] Gibbons RJ, Abrams J, Chatterjee K, Daley J, Deedwania PC, Douglas JS, Ferguson TB Jr, Fihn SD, Fraker TD Jr, Gardin JM, O'Rourke RA, Pasternak RC, Williams SV; American College of Cardiology; American Heart Association Task Force on practice guidelines (Committee on the Management of Patients With Chronic Stable Angina). ACC/AHA 2002 guideline update for the management of patients with chronic stable angina--summary article: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines (Committee on the Management of Patients With Chronic Stable Angina). J Am Coll Cardiol. 2003 Jan 1;41(1):159-68. doi: 10.1016/s0735-1097(02)02848-6. No abstract available. PMID 12570960
- [Background] Saunders JT, Nambi V, de Lemos JA, Chambless LE, Virani SS, Boerwinkle E, Hoogeveen RC, Liu X, Astor BC, Mosley TH, Folsom AR, Heiss G, Coresh J, Ballantyne CM. Cardiac troponin T measured by a highly sensitive assay predicts coronary heart disease, heart failure, and mortality in the Atherosclerosis Risk in Communities Study. Circulation. 2011 Apr 5;123(13):1367-76. doi: 10.1161/CIRCULATIONAHA.110.005264. Epub 2011 Mar 21. PMID 21422391
- [Background] Hallen J, Johansen OE, Birkeland KI, Gullestad L, Aakhus S, Endresen K, Tjora S, Jaffe AS, Atar D. Determinants and prognostic implications of cardiac troponin T measured by a sensitive assay in type 2 diabetes mellitus. Cardiovasc Diabetol. 2010 Sep 15;9:52. doi: 10.1186/1475-2840-9-52. PMID 20843304
- [Background] Fornengo P, Bosio A, Epifani G, Pallisco O, Mancuso A, Pascale C. Prevalence of silent myocardial ischaemia in new-onset middle-aged Type 2 diabetic patients without other cardiovascular risk factors. Diabet Med. 2006 Jul;23(7):775-9. doi: 10.1111/j.1464-5491.2006.01910.x. PMID 16842483
- [Background] Sprague RS, Ellsworth ML. Vascular disease in pre-diabetes: new insights derived from systems biology. Mo Med. 2010 Jul-Aug;107(4):265-9. PMID 20806839
- [Background] Singleton JR, Smith AG, Russell JW, Feldman EL. Microvascular complications of impaired glucose tolerance. Diabetes. 2003 Dec;52(12):2867-73. doi: 10.2337/diabetes.52.12.2867. PMID 14633845
- [Background] Ziegler D, Rathmann W, Dickhaus T, Meisinger C, Mielck A; KORA Study Group. Prevalence of polyneuropathy in pre-diabetes and diabetes is associated with abdominal obesity and macroangiopathy: the MONICA/KORA Augsburg Surveys S2 and S3. Diabetes Care. 2008 Mar;31(3):464-9. doi: 10.2337/dc07-1796. Epub 2007 Nov 26. PMID 18039804
- [Background] Aranda JM Jr, Hill J. Cardiac transplant vasculopathy. Chest. 2000 Dec;118(6):1792-800. doi: 10.1378/chest.118.6.1792. PMID 11115475
- [Background] Omland T, de Lemos JA, Sabatine MS, Christophi CA, Rice MM, Jablonski KA, Tjora S, Domanski MJ, Gersh BJ, Rouleau JL, Pfeffer MA, Braunwald E; Prevention of Events with Angiotensin Converting Enzyme Inhibition (PEACE) Trial Investigators. A sensitive cardiac troponin T assay in stable coronary artery disease. N Engl J Med. 2009 Dec 24;361(26):2538-47. doi: 10.1056/NEJMoa0805299. Epub 2009 Nov 25. PMID 19940289
- [Background] Latini R, Masson S, Anand IS, Missov E, Carlson M, Vago T, Angelici L, Barlera S, Parrinello G, Maggioni AP, Tognoni G, Cohn JN; Val-HeFT Investigators. Prognostic value of very low plasma concentrations of troponin T in patients with stable chronic heart failure. Circulation. 2007 Sep 11;116(11):1242-9. doi: 10.1161/CIRCULATIONAHA.106.655076. Epub 2007 Aug 13. PMID 17698733
- [Background] Rubin J, Matsushita K, Ballantyne CM, Hoogeveen R, Coresh J, Selvin E. Chronic hyperglycemia and subclinical myocardial injury. J Am Coll Cardiol. 2012 Jan 31;59(5):484-9. doi: 10.1016/j.jacc.2011.10.875. PMID 22281251
- [Background] de Lemos JA, Drazner MH, Omland T, Ayers CR, Khera A, Rohatgi A, Hashim I, Berry JD, Das SR, Morrow DA, McGuire DK. Association of troponin T detected with a highly sensitive assay and cardiac structure and mortality risk in the general population. JAMA. 2010 Dec 8;304(22):2503-12. doi: 10.1001/jama.2010.1768. PMID 21139111
- [Background] deFilippi CR, de Lemos JA, Christenson RH, Gottdiener JS, Kop WJ, Zhan M, Seliger SL. Association of serial measures of cardiac troponin T using a sensitive assay with incident heart failure and cardiovascular mortality in older adults. JAMA. 2010 Dec 8;304(22):2494-502. doi: 10.1001/jama.2010.1708. Epub 2010 Nov 15. PMID 21078811
- [Background] Nadir MA, Rekhraj S, Wei L, Lim TK, Davidson J, MacDonald TM, Lang CC, Dow E, Struthers AD. Improving the primary prevention of cardiovascular events by using biomarkers to identify individuals with silent heart disease. J Am Coll Cardiol. 2012 Sep 11;60(11):960-8. doi: 10.1016/j.jacc.2012.04.049. Epub 2012 Aug 22. PMID 22921971
- [Background] Stone PH, Chaitman BR, Stocke K, Sano J, DeVault A, Koch GG. The anti-ischemic mechanism of action of ranolazine in stable ischemic heart disease. J Am Coll Cardiol. 2010 Sep 14;56(12):934-42. doi: 10.1016/j.jacc.2010.04.042. PMID 20828645
- [Background] Deshmukh SH, Patel SR, Pinassi E, Mindrescu C, Hermance EV, Infantino MN, Coppola JT, Staniloae CS. Ranolazine improves endothelial function in patients with stable coronary artery disease. Coron Artery Dis. 2009 Aug;20(5):343-7. doi: 10.1097/MCA.0b013e32832a198b. PMID 19444092
- [Background] Kosiborod M, Arnold SV, Spertus JA, McGuire DK, Li Y, Yue P, Ben-Yehuda O, Katz A, Jones PG, Olmsted A, Belardinelli L, Chaitman BR. Evaluation of ranolazine in patients with type 2 diabetes mellitus and chronic stable angina: results from the TERISA randomized clinical trial (Type 2 Diabetes Evaluation of Ranolazine in Subjects With Chronic Stable Angina). J Am Coll Cardiol. 2013 May 21;61(20):2038-45. doi: 10.1016/j.jacc.2013.02.011. Epub 2013 Mar 10. PMID 23500237
- [Background] Gilead Sciences, Inc. Ranolazine Investigator's Brochure. Section 3.2.2 Placebo Tablets, 30 Mar 2012.
- [Background] FDA drug label for Ranolazine (Ranexa). Accessed via FDA website on 05 October 2012. Last revision Dec 2011. Reference ID: 3164047.